CLINICAL TRIAL: NCT03688724
Title: Perioperative Diaphragm Point-of-care Ultrasound (D-POCUS) for the Detection of Blockage and the Prediction of Postoperative Ventilatory Failure in Patients Who Received Brachial Plexus Blockages Above the Clavicle
Brief Title: Perioperative Diaphragm Point of Care Ultrasound
Acronym: DPOCUS
Status: Completed | Type: Observational
Sponsor: Hospital General Universitario de Valencia (Other)
Responsible Party: Principal Investigator, Lucas Rovira, Principal Investigator, Hospital General Universitario de Valencia
Other Study IDs: ROV-DPOCUS-2018-01
Record Dates: First submitted 2018-09-14; First posted 2018-09-28 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Postoperative Pulmonary Complications; Diaphragm; Brachial Plexus Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is a prospective observational study of a cohort of patients who underwent brachial plexus blockage above the clavicle, and in which diaphragmatic function is observed in both hemidiaphragms by ultrasound (using Diaphragm Thickening Fraction), which allows to obtain the real incidence of Hemidiaphragm palsy in these patients, and estimate the perioperative evolution of both hemidiaphragms.

Hemidiaphragm palsy after brachial plexus block above the clavicle (BPBAC) is frequent, but few patients develop postoperative pulmonary complications (PPC). Little attention has been paid to the contralateral hemidiaphragm as part of the global diaphragmatic function. After BPBAC, global diaphragm function reduces due to ipsilateral hemidiaphragm reduction, but less than expected due to the increase in the contralateral hemidiaphragm function. As a part of the diaphragm function, the contralateral hemidiaphragm function plays a relevant role in the appearance of PPC.

DETAILED DESCRIPTION:
INTRODUCTION Shoulder surgery is known to be a particularly painful stimulus. Perioperative analgesia using brachial plexus block by injection above the clavicle (BPBAC) for shoulder surgery is the standard of care 1,2.

Up to date, ipsilateral diaphragmatic paresis after BPBAC is still very frequent, but few patients develop postoperative pulmonary complications (PPC), and most of them are mild8. There is much concern in avoiding ipsilateral hemidiaphragmatic paralysis to reduce PPC. Little attention has been paid to the contralateral diaphragm and the global diaphragmatic function formed by both hemidiaphragms (the ipsilateral and the contralateral to the BPBAC).

A meticulous study of perioperative diaphragm evolution is needed to answer why some patients after BPBAC develop PPC and others do not.

OUTCOMES The primary objective was to examine the evolution of perioperative hemidiaphragm function with ultrasound (ipsilateral and contralateral) when using BPBAC following shoulder surgery.

the hypothesis is that despite frequent acute ipsilateral hemidiaphragm paralysis after BPBAC, the contralateral hemidiaphragm function increases and preserves global diaphragmatic function in most patients.

METHODS A prospective observational cohort study evaluating perioperative (preoperative and postoperative) diaphragm point-of-care ultrasound (D-POCUS) at an academic tertiary hospital in Spain. Adults undergoing shoulder surgery with planned BPBAC (ISB or SCB) will be eligible for inclusion. Patients planned for not receive BPBAC for any reason will be exclude.

Thickening diaphragm fraction (TF) and diaphragm excursion (DE) were measured in both hemidiaphragms before BPBAC (at the preoperative time) and within 30 min after surgery (at the postoperative time, at least 1 hour after BPBAC).

All measures will be repeated three times in each patient and by the same member of the research team to reduce intra-observer and inter-observer variability. In addition, he will be blinded to the side on which the BPBAC will be performed.

TF was calculated using the following formula: TF = (Tdi-Tde)/Tde x100 (%). TF ipsilateral was the TF measured in the hemidiaphragm ipsilateral to the BPBAC. TF contralateral was the TF measured in the hemidiaphragm contralateral to the BPBAC. TFglobal was the sum of both hemidiaphragm TF to reflect the global diaphragm function. It was calculated using the following formula: (TF Global = (TF ipsilateral + TF contralateral). DE was measured in mm.

Baseline characteristics of participants were collected, including age, gender, comorbidities, respiratory rate (RR), basal SpO2 (Oxygen saturation measured by pulse oximeter), respiratory symptoms, and ARISCAT scale . also data were collect during perioperative, related to BPBAC (loco-regional technique, local anesthetic, concentration, volume of injection); related to intraoperative management (hypnotics, morphic and blocking neuromuscular agents used); and related to postoperative (Train-Of-Four(TOF) scale, visual analog scale (VAS) Pain, RR, SpO2, fraction of inspired oxygen (FiO2), SpO2/FiO2, existence of postoperative pulmonary complications (PPC) ). PPC is defined as the occurrence of dyspnea, tachypnea (RR >20% of preoperative RR), SpO2 <90%, or SpO2/FiO2 <315.

Statistical Analyses Continuous variables will be reported as medians with their interquartile range [IQR] or means with standard deviations (SD) where applicable, and categorical variables as counts and percentages. Group comparisons of continuous variables will be made using the Student t-test or Mann-Whitney U test, or Wilcoxon rank-sum test as appropriate. Chi-square test, Fisher exact test, and Kruskal-Wallis test will be used where appropriate for categorical variables. Analyses will be performed using IBM SPSS Statistics for Windows, Version 24.0 (IBM Corp, Armonk, NY).

SAMPLE SIZE

The sample size was calculated using Gpower 3.1. An effect size of 0.48 was calculated based on the difference between two dependent means (matched pairs) obtained on previous pilot study data. The occurrence of TFcontralateral variation before and after BPBAC was 12±30. A sample size of 59 patients was required to detect a 20% of TFcontralateral variation with 95% power and a two-sided alpha of 0.05. an increase of 10% on sample size was applied.

TOTAL n= 65 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for any type of surgery that requires a supraclavicular or interscalene block.

Exclusion Criteria:

* Age <18 years
* No locoregional blockade over the clavicular for any reason, allergy to local anesthetics, coagulopathy, clinical reason.
* Rejection to enter the observational study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for upper limb surgery
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Contralateral Diaphragm function change | day of surgery (1 hour before surgery starts and 1 hour after surgery ends)
  Thickening fraction (%) change of contralateral hemidiaphragm Before-After Brachial plexus Block

SECONDARY OUTCOMES:
Ipsilateral Diaphragm function change | day of surgery (1hour before surgery starts and 1hour after surgery ends)
  Thickening fraction (%) of ipsilateral hemidiaphragm to BPBAC
Incidence of Postoperative Pulmonary Complications | postoperative 30 min after surgery at PACU(post anesthesia care unit)
  we consider PPC (Dyspnea, oxygen saturation below 92%,PO2/FiO2<300, need for reintubation, high respiratory rate>22)
Incidence of contralateral hemidiaphragm increase after BPBAC. | POSTOPERATIVE 30 min after surgery at PACU (post anesthesia care unit)
  we consider Contralateral hemidiaphragm increase any Thickening Fraction at postoperative >Thickening Fraction at preoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Lucas Rovira, PhD, Principal Investigator — HGUV
Locations (1):
- Hospital General Universitario de Valencia, Valencia, Spain